CLINICAL TRIAL: NCT03341676
Title: Spectroscopic and Diffusion Weighted Analysis of the Effects of Dexamethasone on High Altitude Cerebral Oedema (HACE)
Acronym: D4H
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI175716
Record Dates: First submitted 2017-03-09; First posted 2017-11-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: High Altitude Cerebral Edema
MeSH Terms: conditions — Altitude Sickness | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, Investigator supervising the visit and the Outcome Assessor will be blinded to the treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): 8ml IV 3.3mg/mL dexamethasone
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): 8ml IV 0.9% w/v saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 3.3 mg/mL solution for injection
  Arms: Dexamethasone
Drug: Placebo — Sodium Chloride 0.9% w/v solution for injection
  Arms: Placebo

SUMMARY:
When the brain detects a drop in oxygen levels in the blood (hypoxia) there is a compensatory increase in blood flow. Acute mountain sickness (AMS) is a cluster of symptoms which commonly occur in those ascending to high altitude and experiencing hypoxia due to increased blood flow and then swelling in the brain. Symptoms include headache, nausea, insomnia and fatigue. The exact mechanisms by which AMS develops remains poorly understood. Dexamethasone has been shown to reduce the risk of developing significant brain swelling in other settings. Therefore we hypothesise that administering low dose Dexamethasone could protect against hypoxia induced cerebral and spinal oedema.

DETAILED DESCRIPTION:
The exact mechanisms by which AMS develops remains poorly understood. Interestingly, brain and spinal cord swelling due to low oxygen levels can also occur in the period following surgery to treat thoracic and abdominal aortic aneurysms, dangerous swellings of the major blood vessel in the body. Therefore, if we find a therapeutic benefit of receiving a dose of Dexamethasone in a controlled, reversible setting of hypoxia, it is possible that this could be useful in the treatment of post-operative hypoxia as well.

Work with MRI imaging has demonstrated reduced measures of water movement in patients suffering from cerebral or spinal ischaemia, due to swelling. Specific water channels in brain cells (astrocytes) are involved in the movement of water, and Dexamethasone has been shown to reduce expression of these channels in animal models. Dexamethasone already plays a role in lowering pressure in the brain in the setting of brain tumours. Although high doses are typically used in this setting, there is evidence that lower doses may be equally effective, especially in patients with less severe swelling.

Subjects will be consented and randomised in the weeks before the actual study.

Before entering the tent, the following data will be collected:

* Lake Louise Acute Mountain Sickness self-assessment questionnaire
* Pulse oximetry
* Non-invasive cardiac monitoring (ECG)
* End tidal CO2
* Venous blood collection (Full blood count, renal function, S100 and GFAP)
* Finger-prick blood collection (Purines)
* Magnetic Resonance Angiography

Non-invasive monitoring will continue every 2 hours at the start of the study and around the time of administration of the study drug. They will continue at less frequent intervals throughout the study period. This includes ECG trace and an AMS self-assessment questionnaire.

Venous sampling will be performed on 5 occasions throughout the study. Finger prick sampling will be done at the same time points

Each subject will have 5 MRI scans during the course of the study.

Subjects will be begin hypoxication 1 hour after entering the tent. They will be returned to normal oxygen levels after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Healthy men and women aged 20-50 years
* Ability to fully understand the requirements of the protocol
* Negative pregnancy
* BMI <30 kg/m2

Exclusion Criteria:

* Recent experience of high altitude: Any subject who has visited high altitudes (defined as 8,000 - 12,000 feet above sea level) within 4 weeks of starting the study.
* Abnormal blood pressure: AHA guidelines state blood pressures ≥140/90 mmHg require medical management. Patients with a blood pressure above these parameters will be excluded.
* Any evidence of systemic infection e.g. respiratory tract infection.
* Any evidence of renal disease (i.e. eGFR <60, as this precludes intravenous contrast required for MRI scan)
* History of Tuberculosis
* History of heart disease
* Conditions including but not limited to: Glaucoma (including family history), ocular herpes simplex (risk of corneal perforation), severe affective disorders (particularly if history of steroid-induced psychosis), epilepsy, peptic ulcer, hypothyroidism, history of steroid myopathy, ulcerative colitis, diverticulitis, recent intestinal anastomoses, thromboembolic disorders or myasthenia gravis.
* Breastfeeding
* Current smoker
* Contraindications for MRI
* Known sensitivity to the study drug and / or it's excipients: History of hypersensitivity to steroids (any preparation).
* Taking pharmaceutical preparations or over the counter medications known to interact with intravenous Dexamethasone.
* Current participation in other interventional research

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Differences in oedematous changes in the brain and spinal cord | 0 hour and 8, 11, 22 and 26 hours post hypoxic insult
  Differences in oedematous changes in the brain and spinal cord as measured by changes in brain and spinal cord MRI imaging

SECONDARY OUTCOMES:
Primary blood brain barrier breakdown in hypoxic cytotoxic oedema | 0 hour and 8, 11, 22 and 26 hours post hypoxic insult
  To assess the role of primary blood brain barrier breakdown in hypoxic cytotoxic oedema as measured by variation in serum markers
Assessing the usefulness of biomarkers of hypoxic cerebral changes. | 0 hour and 8, 11, 22 and 26 hours post hypoxic insult
  Change in glial specific (GFAP) and non-glial specific (purines) serum biomarkers from baseline and at 8, 11, 22 and 26 hours post hypoxic insult
Spinal cord model | 0 hour and 8, 11, 22 and 26 hours post hypoxic insult
  To develop a hypoxic spinal cord model for use in future research looking into complex vascular surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Imray, PhD MBBS, Principal Investigator — University Hospital Coventry and Warwickshire NHS Trust
Locations (1):
- University Hospitals Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Fisher O, Benson RA, Wayte S, Kimani PK, Hutchinson C, Imray CHE. Multimodal analysis of the effects of dexamethasone on high-altitude cerebral oedema: protocol for a pilot study. Trials. 2019 Oct 24;20(1):604. doi: 10.1186/s13063-019-3681-0. PMID 31651350